CLINICAL TRIAL: NCT07174999
Title: Prospective Observational Study for Nutritional Evaluation of Infants Receiving Amino Acid-Based Formula at Assiut University Children's Hospital
Brief Title: Nutritional Evaluation of Infants Receiving Amino Acid-Based Formula
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Emeel Fahmy Abd Elmalak, Pediatric Resident, Assiut University
Other Study IDs: AA-Formula-Study-2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cow's Milk Protein Allergy Protein Intolerance Failure to Thrive
Keywords: Amino Acid-Based Formula Infant Nutrition Growth Assessment Food Allergy Nutritional Evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Infants receiving amino acid-based formula who are evaluated at the Nutrition and Gastroenterology Departments, Assiut University Children's Hospital.

SUMMARY:
This study aims to evaluate the growth parameters and nutritional status of infants who are receiving amino acid-based formula due to cow's milk protein allergy or other medical indications.

DETAILED DESCRIPTION:
This prospective observational study will assess infants who are exclusively fed amino acid-based formula. Participants will be followed over a period of 6 months, and anthropometric measurements (weight, length, head circumference) will be recorded monthly. Growth velocity and nutritional status will be analyzed and compared with WHO growth standards.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 1 to 12 months at the time of enrollment.
2. Infants who are exclusevel or predominantly fed amino acid-based formula (AAF) in addition to elimination diet for at least 12 consecutive weeks.
3. Infants who are diagnosed as CMPA by CoMiSS score ≥ 10 and confirmed by OFC test.
4. Infants with informed parental or guardian consent to participate in the study.

Exclusion Criteria:

* 1- Infants with congenital anomalies or syndromes affecting growth and development (e.g., trisomy 21, major cardiac defects).

  2- Infants with chronic systemic illnesses unrelated to feeding (e.g., cystic fibrosis, chronic kidney disease).

  3- Infants receiving additional specialized nutrition support (e.g., parenteral nutrition or tube feeding not involving AAF).

  4- Infants with incomplete or insufficient medical records at the time of assessment.5- Infants who have been on AAF for less than 4 weeks or whose feeding regimen is not stable.

  6- Infants whose parents or legal guardians decline or withdraw informed consent.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include infants aged 1 to 12 months who are exclusively or predominantly receiving amino acid-based formula (AAF) as part of their routine medical care due to established clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean anthropometric z-scores (WAZ, LAZ, WLZ) | Single assessment at enrollment.
  Mean weight-for-age, length-for-age, and weight-for-length z-scores for the study population compared to WHO reference.
Weight-for-Age Z-score (WAZ) - prevalence of underweight | Single assessment at enrollment.
  Prevalence of underweight (weight-for-age z-score < -2) among infants receiving amino acid-based formula, calculated according to WHO growth standards.
Nutritional Status (Weight-for-Age Z-sco | At the time of enrollment (single assessment).
  Assessment of weight-for-age z-score in infants receiving amino acid-based formula compared to WHO growth standards.

SECONDARY OUTCOMES:
Length-for-Age Z-score | At the time of enrollment.
  Measurement of length-for-age z-score according to WHO growth standards.
Head Circumference-for-Age Z-score | At the time of enrollment.
  Measurement of head circumference-for-age z-score according to WHO growth standards.
Gastrointestinal Symptoms | At the time of enrollment (parental report).
  Assessment of gastrointestinal tolerance including vomiting, diarrhea, and constipation

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Ibrahim Hassan, prof, Principal Investigator — Assiut University; Osama Mahmoud Elasheer, prof, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiocchi A, Brozek J, Schunemann H, Bahna SL, von Berg A, Beyer K, Bozzola M, Bradsher J, Compalati E, Ebisawa M, Guzman MA, Li H, Heine RG, Keith P, Lack G, Landi M, Martelli A, Rance F, Sampson H, Stein A, Terracciano L, Vieths S. World Allergy Organization (WAO) Diagnosis and Rationale for Action against Cow's Milk Allergy (DRACMA) Guidelines. World Allergy Organ J. 2010 Apr;3(4):57-161. doi: 10.1097/WOX.0b013e3181defeb9. Epub 2010 Apr 23. No abstract available. PMID 23268426
- [Background] Koletzko S, Niggemann B, Arato A, Dias JA, Heuschkel R, Husby S, Mearin ML, Papadopoulou A, Ruemmele FM, Staiano A, Schappi MG, Vandenplas Y; European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Diagnostic approach and management of cow's-milk protein allergy in infants and children: ESPGHAN GI Committee practical guidelines. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):221-9. doi: 10.1097/MPG.0b013e31825c9482. PMID 22569527